CLINICAL TRIAL: NCT04157530
Title: Clinical Evaluation of Acupuncture in Treating Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH106-REC2-161
Record Dates: First submitted 2018-03-12; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Glaucoma; Acupuncture
MeSH Terms: conditions — Glaucoma | interventions — Acupuncture Therapy; Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sham group (Sham Comparator): 15 subjects with seeds of wang-bu-liu-xing applied on the surface of Jinming and Qiuhou acupoints
  Interventions: Device: wang-bu-liu-xing
- acupuncture group (Experimental): 15 subjects with acupuncture applied to Qingming and Qiuhou with Der-qi
  Interventions: Device: acupuncture
- Electroacupuncture group (Experimental): 15 subjects wth acupuncture, but the needles of Qinming and Qiuhou connected to the electroacupuncture machine after Der-qi
  Interventions: Device: Electroacupuncture

INTERVENTIONS:
Device: wang-bu-liu-xing — wang-bu-liu-xing applied on the surface of Jinming and Qiuhou acupoints
  Other Names: Canon Pneumotonometer
  Arms: sham group
Device: acupuncture — acupuncture applied to Qingming and Qiuhou with Der-qi
  Arms: acupuncture group
Device: Electroacupuncture — acupuncture, but the needles of Qinming and Qiuhou connected to the electroacupuncture machine after Der-qi, the frequencies of stimulus were 6 Hz, the intensity of stimulus was minimal visible muscle twitch
  Arms: Electroacupuncture group

SUMMARY:
The present study predicts that acupuncture or electroacupuncture can reduce intraocular pressure and also can improve quality of life in patients with glaucoma.

DETAILED DESCRIPTION:
Glaucoma is a syndrome, and that is results from intraocular pressure increases cause visual field narrow and blindness. The incidence of adult blindness induced by glaucoma is second in the ophthalmologic disease in the world. Many studies report that both blood circulation in the eye surroundings and intraocular pressure increase play an important role in glaucoma. Several studies show that acupuncture can modulate intraocular pressure and improve activity of central visual acuity and also increase blood flow of eye fundus. Jingming (BL1) can communicate yi and yang, and nourish and clear eyes, Qiuhou (EX-HN7) can transport qi and activate blood, and freely flowing meridian and clear eyes. Therefore, the purpose of the present study was to investigate the therapeutic effect of acupuncture at Jinming and Qiuhou on intraocular pressure in patients with glaucoma. The study designed as a single-blinded, randomized, controlled clinical trial, a total of45 patients with glaucoma divided into three groups, each group was15 subjects as follows: 1) sham group, using the seeds of wang-bu-liu-xing applied on the surface of Jinming and Qiuhou acupoints, one times/day, and each time was 20 min, twice/week for 2 weeks; 2) acupuncture group, the methods were identical to the sham group, but used acupuncture applied to Qingming and Qiuhou with Der-qi; 3) Electroacupuncture group, the methods were identical to acupuncture, but the needles of Qinming and Qiuhou connected to the electroacupuncture machine after Der-qi, the frequencies of stimulus were 6 Hz, the intensity of stimulus was minimal visible muscle twitch. Primary outcome measure was the changes of intraocular pressure, and the second outcome measure was the score changes of WHOQOL-REF (Taiwan version).

The present study predicts that acupuncture or electroacupuncture can reduce intraocular pressure and also can improve quality of life in patients with glaucoma.

ELIGIBILITY:
Inclusion Criteria:

1. Glaucoma for at least three months
2. Do not use ocular hypotensive drugs or use only one ocular hypotensive drug.
3. It is over 20 years old.
4. Men and women are informal.
5. There is no evidence other than glaucoma that shows other eye diseases.
6. Be aware and fill out the consent form yourself.

Exclusion Criteria:

1. Combines other chronic diseases, taking multiple medications such as high blood pressure, diabetes, etc.
2. Those who have had glaucoma surgery.
3. Those who had undergone myopia laser surgery.
4. Can not accept acupuncture points stimulators.
5. Allergic to acupuncture needles.
6. Has a mental illness or is unable to cooperate with the researcher.
7. Do not sign consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
intraocular pressure | 20 min, twice/week for 2 weeks
  Primary outcome measure was the changes of intraocular pressure,

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Liang Hsieh, PhD, Principal Investigator — China Medical University, China
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mac Nair CE, Nickells RW. Neuroinflammation in Glaucoma and Optic Nerve Damage. Prog Mol Biol Transl Sci. 2015;134:343-63. doi: 10.1016/bs.pmbts.2015.06.010. Epub 2015 Jul 10. PMID 26310164
- [Derived] Chen SY, Yieh FS, Liao WL, Li TC, Hsieh CL. Effect of Acupuncture on Intraocular Pressure in Glaucoma Patients: A Single-Blinded, Randomized, Controlled Trial. Evid Based Complement Alternat Med. 2020 Apr 28;2020:7208081. doi: 10.1155/2020/7208081. eCollection 2020. PMID 32419820